CLINICAL TRIAL: NCT00003523
Title: Evaluation of Aminocamptothecin (9-AC, NSC #603071) in Recurrent, Platinum Resistant and Refractory Ovarian Cancer and Primary Peritoneal Carcinoma
Brief Title: Aminocamptothecin in Treating Patients With Recurrent or Refractory Ovarian Epithelial Cancer or Primary Cancer of the Peritoneum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066567; GOG-126I
Record Dates: First submitted 2000-09-11; First posted 2004-05-24 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2005-06

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Drug: aminocamptothecin colloidal dispersion

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminocamptothecin in treating patients with recurrent or refractory ovarian epithelial cancer or primary cancer of the peritoneum.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the antitumor activity of aminocamptothecin colloidal dispersion in patients with platinum-resistant recurrent or refractory ovarian cancer or primary peritoneal carcinoma who have failed on higher priority treatment protocols. II. Determine the nature and degree of toxicity of aminocamptothecin colloidal dispersion in this patient population.

OUTLINE: Patients receive aminocamptothecin colloidal dispersion IV over 120 hours weekly for two of every three weeks. Courses are repeated every 21 days in the absence of disease progression or unacceptable toxicity. Patients are followed every 3 months for 2 years, then every 6 months for 3 years.

PROJECTED ACCRUAL: Approximately 23-56 patients will be accrued for this study within 5-12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent or persistent ovarian epithelial cancer or primary peritoneal carcinoma Progressive disease on platinum-based treatment alone or in combination Two prior treatment regimens allowed only if other regimen was paclitaxel OR recurrence within 6 months of chemotherapy Measurable disease Not eligible for a higher priority GOG protocol

PATIENT CHARACTERISTICS: Age: 13 and over Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT/SGPT no greater than 2.5 times upper limit of normal (ULN) Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL Other: No significant infection Not pregnant Fertile patients must use effective contraception At least 5 years since prior malignancy; no prior chemotherapy or radiotherapy for that malignancy No concurrent malignancy other than non-melanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered No prior treatment with aminocamptothecin Endocrine therapy: At least 4 weeks since prior endocrine therapy Radiotherapy: At least 4 weeks since prior radiotherapy and recovered No prior radiotherapy to site(s) of measurable disease used on this trial No prior radiotherapy to more than 25% of marrow-bearing areas Surgery: At least 4 weeks since prior surgery

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David S. Miller, MD, Study Chair — Simmons Cancer Center
Locations (65):
- United States (64):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Medicine Branch, Bethesda, Maryland
  - Radiation Oncology Branch, Bethesda, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - CCOP - Sooner State, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Miller DS, Blessing JA, Waggoner S, Schilder J, Sorosky J, Bloss J, Schilder R. Phase II evaluation of 9-aminocamptothecin (9-AC, NSC #603071) in platinum-resistant ovarian and primary peritoneal carcinoma: a Gynecologic Oncology Group Study. Gynecol Oncol. 2005 Jan;96(1):67-71. doi: 10.1016/j.ygyno.2004.09.015. PMID 15589582